CLINICAL TRIAL: NCT06029153
Title: Efficacy and Safety of Middle Meningeal Artery Embolization for Treatment of Intractable Migraine： a Single-arm, Self-control, Open-label, Single-center Trial
Brief Title: Efficacy and Safety of Middle Meningeal Artery Embolization for Treatment of Intractable Migraine
Acronym: FAST-EM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Zeguang Ren, Dr., The Affiliated Hospital Of Guizhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAST-EM
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-05

CONDITIONS: Migraine
Keywords: Migraine; Middle meningeal artery; Embolization
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Self-control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Middle meningeal artery embolization (Experimental): Middle meningeal artery embolization with coil.
  Interventions: Procedure: Middle meningeal artery embolization

INTERVENTIONS:
Procedure: Middle meningeal artery embolization — Middle meningeal artery embolization with coil.

SUMMARY:
This study is a single-arm, self-controlled clinical trial that explores and evaluates the efficacy of middle meningeal artery embolization with coil in improving migraine symptoms. The main objectives of the study are to evaluate the effectiveness and safety of the treatment.

DETAILED DESCRIPTION:
This study is a single-arm, self-controlled, open-label, single-center clinical trial that explores and evaluates the efficacy of middle meningeal artery embolization with coil in improving migraine symptoms. The inclusion criteria consist of patients with or without aura migraines, who have experienced persistent, chronic migraines for at least 3 months before screening, and have shown resistance to at least two or more drug treatments, with unsatisfactory therapeutic effects, intolerable side effects, or contraindications. The main objectives of the study are to evaluate the effectiveness and safety of the treatment.

ELIGIBILITY:
Inclusion criteria：

1. Voluntary written informed consent.
2. Age 18~80 years old (inclusive), regardless of gender.
3. Migraine was diagnosed by clinicians, according to The International Classification of Headache Disorders,3rd Edition
4. Patients with intractable migraine or refractory headache with migraine duration of more than 3 months and recurring migraine in the past 90 days before screening.
5. Patients who take two or more drugs are not satisfied with the therapeutic effect, the side effects of drug treatment are difficult to tolerate or have contraindications.
6. Headache frequency should be confirmed within 30 days before screening.
7. Patients with good compliance, willing and able to follow the requirements of treatment and follow-up observation.

Exclusion criteria：

1. Patients with cervical spondylosis and secondary headaches such as otogenic, nasal, and odontogenic patients with a history of trigeminal autonomic headache, other definite causes of headache, or secondary headache.
2. Patients without suitable vascular access.
3. Patients scheduled for surgery within 90 days.
4. The life expectancy of patients is less than 12 months.
5. History of contrast agent allergy.
6. Lactating or pregnant women, or patients with a fertility plan within 1 year.
7. The clinical status of the patient was extremely poor, with an mRS Score ≥4.
8. Participants who had participated in clinical studies of other drugs or medical devices before enrollment and did not meet the primary study endpoint time limit.
9. The investigator judged that the patient had poor compliance and could not complete the study as required.
10. The patient had a clear history of allergies to embolic materials such as Nitinol alloy, cobalt-based alloy, and platinum-tungsten alloy.
11. Patient was allergic to the contrast agent.
12. Patients with other diseases limit their participation in the study, cannot follow up, or affect the scientific integrity of the study.
13. Patients have clotting disorders or are on anticoagulant therapy.
14. Patients have a history of opioid addiction.
15. Researchers believe that patients who are not suitable to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Headache attack frequency (times / month and Headache duration） | At baseline, 90 days after treatment
  Record of headache attack frequency (times / month and Headache duration）

SECONDARY OUTCOMES:
Headache attack frequency (days / month) | At baseline,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  Record of headache attack frequency (days / month)
Days of medication in acute phase and dosage | At baseline,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  Record of days of medication in acute phase and dosage
Severity of headache:Visual Analogue Scale | At baseline,36 hours,day of discharge,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  The scale is mainly composed of a 10cm straight line, one end represents 0 (no pain at al), and the other end represents 10(the worst pain)
Severity of headache:Numerical Rating Scale | At baseline,36 hours,day of discharge,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  The headache level is rated from 0 (no pain) to 10 (the most severe)
Headache aura(nausea,photophobia,phonophobia) frequency | At baseline,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  Record of headache aura
Migraine Disability Assessment | At baseline,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  The Migraine Disability Assessment questionnaire (MIDAS)
Headache Impact | At baseline,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  Headache Impact Test (HIT-6)
Migraine-Specific Questionnaire | At baseline,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  Migraine-Specific Questionnaire（MSQ）
Hospital Anxiety and Depression | At baseline,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  Hospital Anxiety and Depression Scale(HADS)
Clinical Global Impression | At baseline,30 days, 60 days, 90 days, 180 days, 1 year after treatment
  Clinical Global Impression(CGI)

CONTACTS AND LOCATIONS:
Overall Officials: Zeguang Ren, MD. PhD., Study Chair — The Affiliated Hospital Of Guizhou Medical University
Locations (1):
- The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No